CLINICAL TRIAL: NCT00114907
Title: Effects of Black Tea on Cardiovascular Disease in the Mauritian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mauritius (Other)
Collaborators: Mauritius Research Council (Other); Cardiac Centre, Pamplemousses (Other); London South Bank University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: TEA; MRC/RUN-0408
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2005-06

CONDITIONS: Cardiac Disease
Keywords: Tea; Oxidative stress markers; cardiovascular disease; polyphenolics; double blind; Ischaemic cardiac disease
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases | interventions — Tea

INTERVENTIONS:
Behavioral: Consumption of black tea

SUMMARY:
It is proposed to investigate the association between consumption of black tea and various selective fasting blood serum and urine biomarkers in a Mauritian population with ischaemic heart diseases. This study, the first of its kind, will provide clinical data on the potential prophylactic propensities of Mauritian black tea against cardiovascular disease, which remains one of the major health threats to the Mauritian population.

DETAILED DESCRIPTION:
OBJECTIVES

Our broad objectives will be to:

* Survey and recruit patients with ischaemic heart diseases in a randomized sample representative of the Mauritian population (ethnicity, gender, age, social and economical status) and record their medical history,
* Collect fasting blood serum and urine at baseline and after supplement of control volume of tea infusion and water from study group and control group respectively,
* Optimize techniques to determine levels of specific biomarkers from above body fluid samples,
* Investigate existing correlation between tea consumption and risk of cardiovascular diseases in Mauritian population

Our specific objectives will be to:

* Select a randomised group of the Mauritian population, with ischaemic heart disease, who has been referred to the Cardiac Centre, Pamplemousses for Angiography and a group of people showing no risk of cardiovascular diseases
* Inform the people about the motives of the study and seek consent from those willing to participate in the study,
* Evaluate the levels of biomarkers of oxidative stress (total cholesterol, LDL, HDL, triglycerides, homocysteine, atrial natriuretic peptides, brain natriuretic peptides, 8-hydroxydeoxyguanosine, isoprostanes, hydroxyeicosatetraenoic acid, products of protein damage, uric acid and glycosylated haemoglobin) from 8-10 hr fasting blood serum and urine at baseline from all participants
* Supply the study group with a control volume of tea infusion and the control group with the same amount of water for a defined period of time followed by a two week wash out period with water.
* Study biomarkers as above from 8-10 hr fasting blood serum and urine in two week intervals during the supplement regime
* Investigate the existing correlation between tea consumption and levels of biomarkers of cardiovascular diseases in a Mauritian sample population.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 years
* Non smokers
* Left ventricular ejection fraction>40%

Exclusion Criteria:

* Alcohol consumption > 4 standard drinks/day
* Postmenopausal women receiving hormone replacement therapy

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2005-06; Study Completion 2005-06

PRIMARY OUTCOMES:
The study will assess the effect of tea consumption on the incidence of cardiovascular diseases

SECONDARY OUTCOMES:
The effect of tea consumption will be evaluated on a number of markers of oxidative stress associated with cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Theeshan Bahorun, PhD, Principal Investigator — University of Mauritius
Locations (1):
- University of Mauritius, Réduit, Mauritius